CLINICAL TRIAL: NCT04903249
Title: Increasing Physical Activity Among Breast Cancer Survivors: Use of the ORBIT Model to Refine and Test a Novel Approach to Exercise Promotion Based on Affect-regulation
Brief Title: A Single Arm Pilot Study to Refine a Novel Approach to Exercise Promotion Based on Affect-regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Courtney J. Stevens, Assistant Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02000934_1; K08CA259632 (NIH)
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Affect-regulated exercise prescription (Experimental): Participants receive instructions to adjust their pace of exercise so that they feel "fairly good" or better (i.e., a rating of +1 or higher on the Feeling Scale) while exercising and to avoid any increases in intensity that promote feeling "fairly bad" or worse. If no intensity of exercise feels at least "fairly good" participants will be told to exercise at an intensity that feels "as positive as possible."
  Interventions: Behavioral: Core Exercise Promotion Intervention

INTERVENTIONS:
Behavioral: Core Exercise Promotion Intervention — Participants are instructed to increase weekly time spent exercising to >90 minutes over 12 weeks. Exercise will be defined as "activities that use large muscle groups, increase heart rate and breathing rate, and are performed intentionally for the purpose of exercise (as opposed to physical activities of daily living, e.g., housework). Participants complete a videoconferencing visit with the study team and are given task and safety related information pertaining to exercise for survivors of cancer. Participants engage in exercise-related goal-setting and action planning and are provided activity trackers to monitor their activity levels over the 12-week study period.

SUMMARY:
The purpose of this study is to refine the use of an affect-regulated exercise prescription for use with survivors of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Within 5 years of completing curative treatment (surgery, chemotherapy, and radiation) for stage 0-III breast cancer
* <60 mins/week moderate-vigorous physical activity with no major changes for the past 6-months
* Own an Android or iPhone smartphone and willing to use the smartphone to complete app-based surveys during assessment periods
* Willing to wear the ActiGraph monitor during assessment periods
* Access to internet to complete REDCap survey assessments

Exclusion Criteria:

* Non-English speaking/not able to read English
* Evidence of major contraindications for exercise (informed by the 2020 Physical Activity Readiness-Questionnaire (PAR-Q)+)
* Currently pregnant
* History of severe mental illness or currently taking mood stabilizing medications (antipsychotics, anticonvulsants, or lithium)
* Evidence of moderate-severe depressive symptoms (indicated by a score ≥10 on Patient Health Questionnaire-8)
* Evidence of moderate-severe cognitive impairment (indicated by a score < 3 on a 6-item cognitive screener)
* Evidence of clinically significant substance use as indicated by a score of ≥2 on the CAGE-AID screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney J Stevens, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Clinic, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevens CJ, Bobak CA, Morrissette KJ, Thompson RC, Lyons KD, Wallace GM, Emerson AJ, Conroy DE, Williams DM, Chamberlin MD, Bruce ML. Exercise That Feels as Good as Possible: Acceptability of an Affect-Based Exercise Prescription Among Stage 0-III Breast Cancer Survivors. Psychooncology. 2025 Aug;34(8):e70225. doi: 10.1002/pon.70225. PMID 40736469

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant signed consent but did not engage in any reach activities and no data was collected for this individual.
Period: Overall Study
Arm/Group | Affect-regulated Exercise Prescription
Started | 37
Received Intervention | 30
Week 2 Follow-up | 30
Week 6 Follow-up | 30
Week 12 Follow-up | 30
Completed | 30
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.81 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Affect-regulated Exercise Prescription Measured Using the Treatment Acceptability and Preferences (TAP) Measure
Description: A 4-item self-report questionnaire used to measure acceptability of the affect-regulated exercise prescription using a Likert scale ranging from 0 (not at all) to 4 (very much). Total scores range from 0 - 16. Higher scores indicate greater acceptability.
Time Frame: 12-weeks follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | 3.31 (.53)

2. Primary Outcome: Percentage of Sample With Valid Accelerometer Data at Baseline
Description: The number of participants with valid accelerometer data out of the total number of participants in the sample at baseline, multiplied by 100%.
Time Frame: Baseline assessment
Population: Two of the N = 37 participants enrolled at baseline withdrew before starting accelerometer data collection. Thus, accelerometer data at baseline are available from N = 35 participants (i.e., the overall number of participants analyzed for this outcome measure).
Measure: Count of Participants; unit: Participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 35
Participants | 33

3. Primary Outcome: Percentage of Sample With Valid Accelerometer Data at 2-weeks Follow-up
Description: The number of participants with valid accelerometer data out of the total number of participants in the sample during the 2-week follow-up assessment, multiplied by 100%.
Time Frame: 2-weeks follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
Participants | 28

4. Primary Outcome: Percentage of Sample With Valid Accelerometer Data at 6-weeks Follow-up
Description: The number of participants with valid accelerometer data out of the total number of participants in the sample during the 6-week follow-up assessment, multiplied by 100%.
Time Frame: 6-weeks follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
Participants | 28

5. Primary Outcome: Percentage of Sample With Valid Accelerometer Data at 12-weeks Follow-up
Description: The number of participants with valid accelerometer data out of the total number of participants in the sample during the 12-week follow-up assessment, multiplied by 100%.
Time Frame: 12-weeks follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
Participants | 28

6. Primary Outcome: Percentage of Ecological Momentary Assessment (EMA) Survey Prompt Completion
Description: The percentage of ecological momentary assessment (EMA) survey prompts completed by participants during the study out of the total number of EMA survey prompts delivered to participants.
Time Frame: Baseline through 12-weeks follow-up assessments
Population: Two of the N = 37 participants enrolled at baseline withdrew before starting EMA data collection. Thus, EMA data at baseline are available from N = 35 participants (i.e., the overall number of participants analyzed for this outcome measure).
Measure: Number; unit: percentage of EMA prompts completed
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 35
percentage of EMA prompts completed | 84.83

7. Primary Outcome: Number of Participants Who Completed the Exit Interview
Description: Semi-structured interview to assess participants' perceptions regarding their experience participating in the study.
Time Frame: 12-weeks follow-up assessment
Population: Participants who completed the exit interview
Measure: Number; unit: participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
participants | 30

8. Secondary Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 12 Weeks Follow-up
Description: The research grade ActiGraph wGT3X-BT model is a valid measure of physical activity intensity and duration among multiple populations, including breast cancer survivors. Minutes of moderate-vigorous physical activity will be collected from the ActiGraph wGT3X-BT every day for 10-days. Average minutes of moderate-vigorous physical activity completed per day of valid wear time will be calculated.
Time Frame: 12-weeks follow-up assessment
Population: Valid wear accelerometer wear time was defined as 5 or more days of 600 minutes wear time at 12-weeks follow-up. N = 28 participants had valid wear time at 12-weeks follow-up, thus N = 28 is the overall number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes of daily MVPA
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 28
minutes of daily MVPA | 32.97 (40.17)

9. Secondary Outcome: Satisfaction With Study Participation as Measured by the Participant Satisfaction Questionnaire
Description: An 8-item self-report questionnaire used to assess participant satisfaction with study participation using a Likert scale ranging from 1 to 4 . Scores are summed and then averaged; total scores range from 1- 4. Higher scores indicate greater satisfaction.
Time Frame: 12-weeks follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | 3.33 (.63)

10. Secondary Outcome: Study Retention at 2-weeks Follow-up
Description: Number of participants who complete the 2-week follow-up assessment out of the number of participants who enroll in the study.
Time Frame: 2-weeks follow-up assessment
Measure: Number; unit: participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
participants | 30

11. Secondary Outcome: Study Retention at 6-weeks Follow-up
Description: Number of participants who complete the 6-week follow-up assessment out of the number of participants who enroll in the study.
Time Frame: 6-weeks follow-up assessment
Measure: Number; unit: participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
participants | 30

12. Secondary Outcome: Study Retention at 12-weeks Follow-up
Description: Number of participants who complete the 12-week follow-up assessment out of the number of participants who enroll in the study.
Time Frame: 12-weeks follow-up assessment
Measure: Number; unit: participants
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
participants | 30

13. Other Pre Specified Outcome: Change Overtime in Cancer-related Fatigue Measured Using the PROMIS Fatigue Short Form 8a
Description: An 8-item self-report measure with response options ranging from 1 (not at all) to 5 (very much) and fatigue interference ranging from 1 (never) to 5 (always) over the past 7 days. Total scores range from 8 - 40. Higher scores reflect more fatigue.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
units on a scale | -1.50 (5.40)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.137, t-test, 2 sided

14. Other Pre Specified Outcome: Change Overtime in Health-related Quality of Life Measured Using the PROMIS Global Health Scale
Description: A 10-item self-report measure with response options ranging from 1 (poor/never/not at all) to 5 (excellent/completely/always) for items 1-9 and 0 (no pain) to 10 (worst pain imaginable) for the item 10. Total scores range from 9 - 45. Higher scores represent better health-related quality of life.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | .60 (3.07)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.293, t-test, 2 sided

15. Other Pre Specified Outcome: Change Overtime in Physical Functioning Measured Using The PROMIS Physical Function Short Form 8a
Description: An 8-item self-report measure with response options ranging from 1 (unable to do) to 5 (without any difficulty) and the degree to which health limits specific activities on a scale from 1 (cannot do) to 5 (not at all). Total scores range from 8 - 40. Higher scores reflect better physical function.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | .40 (4.24)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.609, t-test, 2 sided

16. Other Pre Specified Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using The Godin Leisure-Time Exercise Questionnaire at 2 Weeks Follow up
Description: The Godin Leisure-Time Exercise Questionnaire is a brief self-report measure that asks participants to report how many minutes they spent participating in moderate and vigorous physical activity on a given day. Participants will report total minutes of moderate-vigorous physical activity completed per day for 10-days. Average minutes of moderate-vigorous physical activity completed per day will be calculated.
Time Frame: 2-weeks follow-up assessment
Population: Data was missing from N = 1 participant, total sample size at 2 weeks follow up was N = 30.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 29
minutes per day | 16.36 (15.04)

17. Other Pre Specified Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using The Godin Leisure-Time Exercise Questionnaire at 6 Weeks Follow up
Description: as for outcome 16
Time Frame: 6-weeks follow-up assessment
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
minutes per day | 11.61 (14.70)

18. Other Pre Specified Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using The Godin Leisure-Time Exercise Questionnaire at 12 Weeks Follow up
Description: as for outcome 16
Time Frame: 12-weeks follow-up assessment
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
minutes per day | 17.13 (16.77)

19. Other Pre Specified Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 2 Weeks Follow-up
Description: as for outcome 8
Time Frame: 2-weeks follow-up assessment
Population: Valid wear accelerometer wear time was defined as 5 or more days of 600 minutes wear time at 2-weeks follow-up. N = 28 participants had valid wear time at 2-weeks follow-up, thus N = 28 is the overall number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes of daily MVPA
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 28
minutes of daily MVPA | 30.48 (17.20)

20. Other Pre Specified Outcome: Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 6 Weeks Follow-up
Description: as for outcome 8
Time Frame: 6-weeks follow-up assessment
Population: Valid wear accelerometer wear time was defined as 5 or more days of 600 minutes wear time at 6-weeks follow-up. N = 28 participants had valid wear time at 6-weeks follow-up, thus N = 28 is the overall number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes of daily MVPA
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 28
minutes of daily MVPA | 29.11 (15.84)

21. Other Pre Specified Outcome: Change in Voluntary Exercise Behavior Measured Using The Voluntary Exercise Questionnaire
Description: A 6-item self-report measure of exercise performed over the last month and week. Two items range from 1 (never) to 7 (often) and four items range from 0 (0 days per week) to 7 (7 days per week). Total scores range from 2-21. Higher scores reflect higher levels of voluntary exercise behavior.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | 1.93 (4.46)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.025, t-test, 2 sided

22. Other Pre Specified Outcome: Change in Physical Activity Category Completed in the Past Month Measured Using the Stanford Leisure-Time Activity Categorical Item (L-Cat)
Description: A single item self-report measure that present six statements describing various levels of monthly physical activity. Response options range from 1 (I did not do much physical activity) to 5 (I did vigorous activities almost daily). Total scores range from 1-5. Higher scores reflect more vigorous, more frequent physical activities completed in the past month.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | .80 (.89)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p < 0.001, t-test, 2 sided

23. Other Pre Specified Outcome: Change in Intentions to Engage in Physical Activity Measured Using The Exercise Intentions Scale
Description: A 5-item self-report measure of intentions to engage in physical activity. Response options range from 1 (not at all likely) to 7 (very likely). Responses are summed and then averaged; total scores range from 1-7. Higher scores represent stronger intentions to engage in physical activity.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | .27 (1.49)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = .327, t-test, 2 sided

24. Other Pre Specified Outcome: Change in Self-efficacy for Exercise Measured Using The Barriers Specific Self-Efficacy for Exercise Scale
Description: A 13-item self-report measure of one's perceived capability to exercise regularly despite commonly identified barriers to participation. Response options range from 0 (not at all confident) to 100 (highly confident). Responses are summed and then averaged; total scores range from 0% - 100%, higher scores represent greater self-efficacy for exercise.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | -2.82 (21.58)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.479, t-test, 2 sided

25. Other Pre Specified Outcome: Change in Intrinsic Motivation for Exercise Measured Using The Behavioral Regulations in Exercise Questionnaire (BREQ-2)
Description: A 4-item self-report scale depicting intrinsic motivation for exercise. Response options range from 0 (not true for me) to 4 (very true for me). Responses are summed and then averaged; total scores range from 0-4. Higher scores indicate greater intrinsic motivation for exercise.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | -.14 (.96)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.424, t-test, 2 sided

26. Other Pre Specified Outcome: Change in Affective Attitudes About Exercise Using The Instrumental and Affective Attitudes About Exercise Scale
Description: A 4-item self-report measure of affective attitudes for exercise. Response options range from -5 to 5. Responses are summed and then averaged; total scores range from -5 to 5. Higher scores more favorable affective attitudes about exercise.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | -.36 (1.78)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.279, t-test, 2 sided

27. Other Pre Specified Outcome: Change in Instrumental Attitudes About Exercise Using The Instrumental and Affective Attitudes About Exercise Scale
Description: A 4-item self-report measure of instrumental attitudes for exercise. Response options range from -5 to 5. Responses are summed and then averaged; total scores range from -5 to 5. Higher scores more favorable instrumental attitudes about exercise.
Time Frame: Baseline and 12-weeks follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affect-regulated Exercise Prescription
Number analyzed (Participants) | 30
score on a scale | -.49 (1.33)
Statistical Analysis 1: Comparison: Affect-regulated Exercise Prescription; Test type: Other; p = 0.052, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 15 weeks. After participants initially enroll in the study there is often a period of a week or more before they can be scheduled for their intervention orientation meeting. The intervention portion of the study last 12 weeks. Often it takes a week or more before participants can be scheduled for their exit interview after the end of the 12 week intervention. Thus, participants are assessed for a period of approximately 15 weeks.
Arm/Group | Affect-regulated Exercise Prescription
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT04903249/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT04903249/ICF_001.pdf